CLINICAL TRIAL: NCT01576757
Title: Harvest, Isolation and Culture of Cardiac Stem Cells From Endomyocardial Biopsies
Status: Withdrawn | Type: Observational
Why Stopped: There were no funds for the study.
Sponsor: University of Louisville (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Roberto Bolli, Endowed Chair Professor, University of Louisville
Other Study IDs: UL-11.0146
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure
Keywords: Stem cell therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy samples are taken at the time of right heart catheterization. They are frozen in a GMP facility at the University of Louisville. The tissue is shipped either to the Institue of Molecular Caridology, Louisville, KY or shipped overnight to the Brigham and Women's Hospital in Boston, MA. The tissue is enzymatically dissociated, and cardiac stem cells are isolated and maintained in culture for 6-8 passages (point of clinical utility). During that time period, experimentation is carried out to charcterize the biological attributes of these cell populations. After this experimentation is complete, the cultures are destroyed in accordance with the biohazard handling policies of the individual institution.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure: Patients with heart failure from any cause will be considered as potential participants given their clinical background meets eligibility criteria.

SUMMARY:
The purpose of this study is to determine whether the harvest, isolation and culture of cardiac stem cells from endomyocardial biopsies is feasible.

DETAILED DESCRIPTION:
Heart failure is a devastating condition affecting nearly 6 million patients in the United States alone. Ischemic cardiomyopathy, or pump failure secondary to previous heart attack, is considered by many to be the leading cause of heart failure. Stem cell therapy, or regeneration of the lost myocardium, is an intervention that has the potential for reversing the detrimental effects of this disease. Recently published evidence has shown preliminary results indicating the safety and feasibility of utilizing cardiac stem cells for the treatment of ischemic cardiomyopathy. The ability to use a commonly practiced method, such as endomyocardial biopsy, to isolate and expand stem cell cultures could, potentially, make this therapy widely available. The results of this study will be important for the design of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Any heart failure patient scheduled for RHC without contraindication for biopsy.
2. Any patient undergoing biopsy for diagnostic purposes may also be included in the study.

Exclusion Criteria:

1. Severe comorbidities (AST, ALT, serum creatinine > 3 times the upper limit of normal).
2. Pregnancy or women of childbearing potential.
3. Anticoagulation which cannot be stopped for 5-7 days.
4. Hepatitis B, C or HIV.
5. Inability to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure undergoing evaluation for medical management at the University of Louisville or Jewish Hospital in Louisville, KY will be considered for participation based on the evaluation of enrollment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of using endomyocardial biopsy samples to isolate and expand cardiac stem cell cultures. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bolli, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States